CLINICAL TRIAL: NCT05174455
Title: Phase II Study of Niraparib for Leiomyosarcoma With Alterations in the Homologous Recombination DNA Repair Pathway
Brief Title: Niraparib for the Treatment of Leiomyosarcoma
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: PI decision
Sponsor: David Liebner, MD (Other)
Responsible Party: Sponsor-Investigator, David Liebner, MD, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSU-21214; NCI-2021-12582 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2021-12-13; First posted 2021-12-30 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Locally Advanced Leiomyosarcoma; Metastatic Leiomyosarcoma; Stage III Retroperitoneal Sarcoma AJCC v8; Stage IIIA Retroperitoneal Sarcoma AJCC v8; Stage IIIB Retroperitoneal Sarcoma AJCC v8; Stage IV Retroperitoneal Sarcoma AJCC v8; Unresectable Leiomyosarcoma
MeSH Terms: conditions — Leiomyosarcoma | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Niraparib) (Experimental): Patients receive niraparib PO QD. Cycles repeat every 28 days for 15 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Niraparib Tosylate Monohydrate

INTERVENTIONS:
Drug: Niraparib Tosylate Monohydrate — Given PO
  Other Names: Zejula

SUMMARY:
This phase II trial tests whether niraparib works to shrink tumor in patients with leiomyosarcoma. Niraparib is an inhibitor of PARP, an enzyme that helps repair deoxyribonucleic acid (DNA) when it becomes damaged. Blocking PARP may help keep cancer cells from repairing their damaged DNA, causing them to die. PARP inhibitors are a type of targeted therapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate whether niraparib tosylate monohydrate (niraparib) shows preliminary evidence of clinical activity among subjects with leiomyosarcoma (LMS) with genomic alterations in the homologous recombination (HR) pathway as measured by the confirmed objective response rate (ORR).

SECONDARY OBJECTIVES:

I. To evaluate the clinical benefit rate (CBR) associated with niraparib treatment in the study population.

II. To evaluate the progression free survival (PFS) associated with niraparib treatment in the study population.

III. To evaluate the overall survival (OS) associated with niraparib treatment in the study population.

IV. To evaluate the overall safety and tolerability of niraparib treatment in the study population.

EXPLORATORY OBJECTIVES:

I. To evaluate predictive biomarkers of response to niraparib. II. To evaluate genomic mechanisms of resistance following treatment benefit with niraparib.

III. To evaluate previous treatment response as a marker of response to niraparib.

OUTLINE:

Patients receive niraparib orally (PO) once daily (QD). Cycles repeat every 28 days for 15 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 5 years or until death.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have histologically documented LMS. Pathology review and confirmation of diagnosis will occur at the site enrolling the patient on this study.
* Patients must have had a recent, within six months of screening, tumor biopsy testing positive for pathogenic mutation or homozygous loss of either BARD1, BRCA1, BRCA2, BRIP1, PALB2, RAD51, RAD51B, RAD51C, or RAD51D using a clinically validated next-generation (NGS) sequencing panel.

  * Variant pathogenicity will be arbitrated by the primary investigative team
* Patients must have locally advanced and unresectable or metastatic disease
* Patients must have disease which is measurable at study entry according to Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1. Additionally, patients must have a site of disease deemed accessible for biopsy at no or minimal risk to the patient (including through the use of image-guidance). If there are questions regarding the feasibility of biopsy, the case should be reviewed with interventional radiology or the appropriate department at the study site
* Patients must have had prior progression on, or intolerance to, at least one line of systemic therapy for advanced LMS. Adjuvant therapy administered after curative resection will not qualify as prior treatment. There is no upper limit on the number of prior therapies received
* Participant must have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Participant must be >= 18 years of age
* Absolute neutrophil count >= 1,500/uL
* Platelets >= 100,000/uL
* Hemoglobin >= 9 g/dL
* Serum creatinine =< 1.5 x upper limit of normal (ULN) or calculated creatinine clearance >= 30 mL/min using the Cockcroft-Gault equation
* Total bilirubin =< 1.5 x ULN (=< 2.0 in patients with known Gilbert's syndrome) OR direct bilirubin =< 1 x ULN
* Aspartate aminotransferase and alanine aminotransferase =< 2.5 x ULN unless liver metastases are present, in which case they must be =< 5 x ULN
* Participant receiving corticosteroids may continue as long as their dose is stable for least 4 weeks prior to initiating protocol therapy
* Female participant has either a negative highly sensitive urine or a serum pregnancy test within 72 hours prior to taking study treatment if of childbearing potential and agrees to abstain from activities that could result in pregnancy from screening through 180 days after the last dose of study treatment, or is of nonchildbearing potential. Nonchildbearing potential is defined as follows (by other than medical reasons):

  * >= 45 years of age and has not had menses for > 1 year
  * Patients who have been amenorrhoeic for < 2 years without history of a hysterectomy and oophorectomy must have a follicle stimulating hormone value in the postmenopausal range upon screening evaluation
  * Post-hysterectomy, post-bilateral oophorectomy, or post-tubal ligation. Documented hysterectomy or oophorectomy must be confirmed with medical records of the actual procedure or confirmed by an ultrasound. Tubal ligation must be confirmed with medical records of the actual procedure, otherwise the patient must be willing to use 2 adequate barrier methods throughout the study, starting with the screening visit through 180 days after the last dose of study treatment. Information must be captured appropriately within the site's source documents. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient.
  * Females on hormone replacement therapy (HRT) and whose menopausal status is in doubt will be required to use one of the non-estrogen hormonal highly effective contraception methods if they wish to continue their HRT during the study. Otherwise, they must discontinue HRT to allow confirmation of postmenopausal status before study enrollment
* Male participant agrees to use an adequate method of contraception starting with the first dose of study treatment through 90 days after the last dose of study treatment. Note: Abstinence is acceptable if this is the established and preferred contraception for the patient
* Participant must be able to understand the study procedures and agree to participate in the study by providing written informed consent
* Participant must have normal blood pressure or adequately treated and controlled hypertension (i.e. systolic blood pressure =< 140 mmHg and diastolic blood pressure =< 90 mmHg).

Exclusion Criteria:

* Patients must not have had any previous treatment with any poly(adenosine diphosphate[ADP]-ribose) polymerase (PARP) inhibitors
* Participant must not be simultaneously enrolled in any interventional clinical trial
* Participant must not have had major surgery =< 4 weeks prior to initiating protocol therapy and participant must have recovered from any surgical effects
* Participant must not have received investigational therapy =< 4 weeks, or within a time interval less than at least 5 half-lives of the investigational agent, whichever is shorter, prior initiating protocol therapy
* Participant receiving non-steroidal anti-estrogen agents must discontinue their use at least two weeks prior to study entry
* Participant has had radiation therapy encompassing > 20% of the bone marrow within 2 weeks; or any radiation therapy within 1 week prior to Day 1 of protocol therapy
* Participant must not have a known hypersensitivity to niraparib components or excipients.
* Participant must not have received a transfusion (platelets or red blood cells) =<4 weeks prior to initiating protocol therapy
* Participant must not have received colony-stimulating factors (e.g., granulocyte colony-stimulating factor, granulocyte macrophage colony-stimulating factor, or recombinant erythropoietin) within 4 weeks prior to initiating protocol therapy
* Participant has had any known Grade 3 or 4 anemia, neutropenia or thrombocytopenia due to prior chemotherapy that persisted > 4 weeks and was related to the most recent treatment
* Participant must not have any known history or current diagnosis of myelodysplastic syndrome (MDS) or acute myeloid leukemia (AML)
* Participant must not have a serious, uncontrolled medical disorder, nonmalignant systemic disease, or active, uncontrolled infection. Examples include, but are not limited to, uncontrolled ventricular arrhythmia, recent (within 90 days) myocardial infarction, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, or any psychiatric disorder that prohibits obtaining informed consent
* Participant must not have had diagnosis, detection, or treatment of another type of cancer =< 2 years prior to initiating protocol therapy (except basal or squamous cell carcinoma of the skin and cervical cancer that has been definitively treated)
* Participant has leptomeningeal disease, carcinomatous meningitis, symptomatic brain metastases, or radiologic signs of central nervous system (CNS) hemorrhage.

  * Note: Participants with asymptomatic brain metastases (i.e. off corticosteroids and anticonvulsants for at least 7 days) are permitted
* Participant has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [qualitative] is detected).
* Prior history of posterior reversible encephalopathy syndrome (PRES)
* History of severe renal impairment
* History of severe liver impairment
* Any clinically significant gastrointestinal (GI) abnormalities that may alter absorption such as malabsorption syndrome or major resection of the stomach and/or bowels.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Confirmed objective response rate (ORR) | Within first 6 months of study treatment
  Defined as complete response + partial response measured by Response Evaluation Criteria in Solid Tumors version 1.1 (RECISTv1.1). Will be calculated as the proportion of patients who achieve a response (complete response + partial response) within the first 6 months of treatment divided by the total number of evaluable patients. An evaluable patient is defined as an eligible patient who has received at least one dose of therapy. All evaluable patients will be included in calculating the ORR for the study along with corresponding 95% binomial confidence intervals (CIs) (assuming that the number of patients who respond is binomially distributed).

SECONDARY OUTCOMES:
Incidence of adverse events (AEs) | Up to 2 years after study treatment
  Frequency and severity of AEs and tolerability of the regimen will be collected and summarized by descriptive statistics. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns. All patients who have received at least one dose of the therapeutic agents will be evaluable for toxicity and tolerability.
Confirmed clinical benefit rate (CBR) | Within first 6 months of study treatment
  Defined as complete response + partial response + stable disease. Will be calculated with 95% binomial CIs.
Progression-free survival (PFS) | From first treatment with the study drug to the earliest of either disease progression or death from any cause, assessed up to 2 years
  Will initially be modeled using Kaplan-Meier methods, resulting in median survival times with 95% CI, assuming sufficient events have occurred.
Overall survival (OS) | From first treatment with the study drug to the death from any cause, assessed up to 2 years
  Will initially be modeled using Kaplan-Meier methods, resulting in median survival times with 95% CI, assuming sufficient events have occurred.

CONTACTS AND LOCATIONS:
Overall Officials: David Liebner, MD, Principal Investigator — Ohio State University Comprehensive Cancer Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: The Jamesline — http://cancer.osu.edu